CLINICAL TRIAL: NCT04237571
Title: Community Agriculture Nutritional Enterprises (CANE) Meal Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dawn Brewer (Other)
Responsible Party: Sponsor-Investigator, Dawn Brewer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 55735
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Diet, Healthy; Life Style, Healthy
Keywords: fruits; vegetables; exercise; community; education
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CANE Adult Participants (Experimental): This sample population consists of an active intervention group of prior Tanglewood to Table walking program adult participants.
  Interventions: Behavioral: CANE Meal Program

INTERVENTIONS:
Behavioral: CANE Meal Program — Participants will be encouraged to pick up a healthy meal from the Community Agriculture Nutritional Experience (CANE) Kitchen in Whitesburg, Kentucky once a week for five weeks. The meals will consist of at least one serving of a fruit or a vegetable. At each meal, education materials will be distributed, including the recipe for the healthy meals and nutrition handouts that are linked to the recipes. Additional information about the ways the nutrients in the meal may help protect from the negative effects of environmental pollutants will be included.

SUMMARY:
Previous adult participants of the Tanglewood to Table walking program will be recruited to enroll in the CANE Meal Program. This program will encourage participants to pick up a healthy meal from the CANE Kitchen each week for five weeks. The meal will consist of at least one serving of fruit or vegetables. At each meal, educational materials will be distributed, including the recipe for healthy meals and nutrition handouts that are linked to the recipes. Additional information about the ways the nutrients in the meal may help protect from the negative effects of environmental pollutants will be included. Surveys, blood pressure, height, weight, waist circumference and carotenoid status will be assessed before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* previous participant in Tanglewood to Table Walking Program

Exclusion Criteria:

* institutionalized adults
* children under the age of 18
* adults with impaired consent capacity
* incarcerated adults

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Change in fruit and vegetable consumption. | Five weeks
  Fruit and vegetable consumption will be assessed with a food frequency questionnaire pre- and post-intervention. This questionnaire asks participants to estimate the frequency of consumption on a ten point scale (from never to three times per day) of 45 specific fruits or vegetables. Aggregate scores range from 0-450 with higher scores indicating increased consumption.
Change in weight. | Five weeks
  Body weight will be measured on a digital scale pre- and post-intervention.
Change in waist circumference | Five weeks
  Waist circumference will be measured with a tape measure pre- and post-intervention.
Change in total blood pressure | Five weeks
  Systolic and diastolic blood pressure will be measured pre- and post-intervention using a digital blood pressure machine.
Change in carotenoid status | Five weeks
  Carotenoid status will be measured via carotenoid RS scanner, an objective measure of diet-derived pigments in the skin.
Change in knowledge of nutrition and environmental pollution. | Five weeks
  Knowledge of nutrition and environmental pollution will be assessed using a mixed 6-item survey containing 4 "yes" "no" "not sure" questions and two multiple choice knowledge questions. The questionnaire does not have an absolute range, but a higher percent of "not sure" responses indicates less knowledge of nutrition and pollution; while a higher percentage of absolutely correct responses indicates increased knowledge. Data will be reported as the change from pre- to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Brewer, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No